CLINICAL TRIAL: NCT03049852
Title: A Phase 2a Multicenter, Randomized, Vehicle-Controlled, Dose Escalating Study to Evaluate the Safety, Efficacy and Pharmacokinetics of CBT-001 Ophthalmic Solution in Patients With Primary or Recurrent Pterygium
Brief Title: Safety and Efficacy of CBT-001 Ophthalmic Solution in Patients With Pterygium
Acronym: Pterygium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cloudbreak Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBT-CS101
Record Dates: First submitted 2017-02-03; First posted 2017-02-10 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2018-09

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CBT-001 Ophthalmic Solution Single dose (Experimental): One drop in the study administered one time only for one day
  Interventions: Drug: CBT-001 single dose
- Vehicle (Placebo Comparator): One drop in the study administered three times daily (TID) for 4 weeks
  Interventions: Drug: Vehicle
- CBT-001 Ophthalmic Solution Multidose (Experimental): One drop in the study administered three times daily (TID) for 4 weeks
  Interventions: Drug: CBT-001 Multi-dose

INTERVENTIONS:
Drug: CBT-001 single dose — One drop in the study administered one time
  Arms: CBT-001 Ophthalmic Solution Single dose
Drug: Vehicle — One drop in the study administered three times daily (TID) for 4 weeks
  Arms: Vehicle
Drug: CBT-001 Multi-dose — One drop in the study administered three times daily (TID) for 4 weeks
  Arms: CBT-001 Ophthalmic Solution Multidose

SUMMARY:
Stage 1: Single Ascending Dose, Safety, Tolerability and Pharmacokinetics (n=24)

Stage 2: Multiple Dose, Safety and Efficacy Study with 28-day Dosing and 5 months Followup (n=51)

DETAILED DESCRIPTION:
Stage 1: Single Ascending Dose, Safety, Tolerability and Pharmacokinetics (n=24)

Objectives are to evaluate ocular safety and tolerability by biomicroscopy, ophthalmoscopy, intraocular pressure and visual acuity, and to assess general safety by physical exams, vital signs, clinical laboratory tests and adverse events reporting and to evaluate systemic CBT-001 exposure by Cmax, Tmax and an estimation of the area under the curve (AUC).

Three dose cohorts will be planned with a dose ascending strategy to guide dose concentrations (n=8 per Cohort x 3 cohorts = 24). Primary pterygium patients will be selected in this phase because the main goal is to assess the safety and tolerability of CBT-001 and primary pterygium patients are much easier to recruit. The ~8 primary pterygium patients from each Cohort will be administered a single ocular drug dose at Day 1 in the eye with primary pterygium; the unaffected eye will be dosed with vehicle. Examinations will be performed at both screening day (Day 0) and Day 1. Blood samples at pre-dose, 0.25, 0.5, 1, 2, 4 and 8 hours post dose will be taken at Day 1 to assess systemic pharmacokinetics (PK). The data will be reviewed by Data Review Committee (DRC) to determine whether to initiate enrollment for the next Cohort.

Cohort 1 will begin at the lowest CBT-001 concentration of 0.02%, followed by an increasing dose to 0.05% for Cohort 2 and then to 0.2% for Cohort 3. If no safety issues are found at all doses, the highest dose of 0.2% will be used for the next phase study.

Stage 2: Multiple Dose, Safety and Efficacy Study with 28-day Dosing and 5 months Followup (n=51)

Objectives are to evaluate ocular and systemic safety of CBT-001 in primary or recurrent patients that have moderate to severe pterygium vascularity and to assess whether CBT-001 is efficacious in reducing pterygium vascularity and pterygium lesion growth. The dosing will be 4 weeks. The followup period will be 5 months.

Study Population Characteristics: Approximately 50 (30 primary pterygium and 20 recurrent) patients will be enrolled at up to 3 centers to have an estimated 40 patients complete the study based on an anticipated dropout rate of 20%. Although we have no evidence to suggest attrition due to Adverse Effects (AEs), the dropout rate is most conservative based on industry experience in comparable clinical studies. Patients will be randomized in a 1:1 treatment allocation to receive either CBT-001 0.2% or Vehicle.

Dosage/Dose regimen: One drop of the assigned study medication will be administered in the study eye TID for 4 weeks. The study eye is defined as the qualified eye (i.e., the eye meeting the inclusion criterion for primary or recurrent pterygium). If both eyes are qualified, then the eye with the more severe vascularity grade on the Pterygium Hyperemia Grading Scale at the baseline (Day 1) visit will be the study eye. If both eyes meet the criterion and have the same severity, the right eye will be the study eye. Patients with bilateral pterygium will administer study medication only in the study eye. The fellow eyes in all study subjects will be untreated.

ELIGIBILITY:
Inclusion Criteria:

* Primary pterygium with moderate vascularity (Pterygium Hyperemia Grading Scale ≥ 3)

Exclusion Criteria:

* Active ocular disease, corneal abnormalities other than pterygium, active ocular infection, or any ocular pathology unrelated to pterygium in either eye that could affect the assessment of the pterygium
* History of ocular herpes disease in either eye
* Any ocular surgical procedure within the last 3 months
* Female patients who are pregnant, nursing, or planning a pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, M.D., Principal Investigator — Harvard Eye Associates
Locations (1):
- Harvard Eye Associates, Laguna Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CBT-001 Ophthalmic Solution Single Dose: CBT-001 Ophthalmic Solution Single dose in one day
- Vehicle Multi-dose; CBT-001 Ophthalmic Solution Multi-dose: One drop in the study administered three times daily (TID) for 4 weeks
Period: Overall Study
Arm/Group | CBT-001 Ophthalmic Solution Single Dose | Vehicle Multi-dose | CBT-001 Ophthalmic Solution Multi-dose
Started | 24 | 25 | 26
Completed | 24 | 24 | 26
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CBT-001 Ophthalmic Solution Single Dose: One drop in the study administered one time
  CBT-001: One drop in the study administered one time
- Vehicle Multi-dose: One drop in the study administered three times daily (TID) for 4 weeks
  Vehicle: One drop in the study administered three times daily (TID) for 4 weeks
- CBT-001 Ophthalmic Solution Multi-dose: One drop in the study administered three times daily (TID) for 4 weeks
  CBT-001: One drop in the study administered three times daily (TID) for 4 weeks
- Total: Total of all reporting groups
Arm/Group | CBT-001 Ophthalmic Solution Single Dose | Vehicle Multi-dose | CBT-001 Ophthalmic Solution Multi-dose | Total
Number analyzed (Participants) | 24 | 25 | 26 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.6) | 49.4 (10.7) | 52.0 (12.1) | 50.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 14 | 38
  Male | 11 | 14 | 12 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 24 | 21 | 24 | 69
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 26 | 75

OUTCOME MEASURES:

1. Primary Outcome: Pterygium Vascularity Change Assessed Using the Pterygium Hyperemia Grading Scale
Description: The primary efficacy variable is the change from baseline (Day 1) in severity grade of pterygium vascularity at Week 4. Pterygium vascularity intensity is based on color coordinates as measured by digital image analysis of pterygium photographs. The quantitative analysis of photographs using a 5-point Pterygium Hyperemia Grading Scale (0 = absent, 1 = trace, 2 = mild, 3 = moderate, 4 = severe) will be conducted at an independent image reading center.
Time Frame: Change from baseline at 4 weeks
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: grade
Groups:
- Vehicle Multi-dose: One drop in the study administered three times daily (TID)
  Vehicle: One drop in the study administered three times daily (TID) for 4 weeks
- CBT-001 Ophthalmic Solution Multi-dose: One drop in the study administered three times daily (TID)
  CBT-001: One drop in the study administered three times daily (TID) for 4 weeks
Arm/Group | Vehicle Multi-dose | CBT-001 Ophthalmic Solution Multi-dose
Number analyzed (Participants) | 23 | 25
grade | 0 (0.5) | -0.8 (0.7)
Statistical Analysis 1: Comparison: Vehicle Multi-dose vs CBT-001 Ophthalmic Solution Multi-dose; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Ocular and General Safety and Tolerability
Description: The ocular safety and tolerability are measured by biomicroscopy, ophthalmoscopy, intraocular pressure and visual acuity, and to assess general safety by physical exams, vital signs, clinical laboratory tests and adverse events reporting
Time Frame: One day
Population: mITT
Measure: Number; unit: participants
Groups:
- CBT-001 Ophthalmic Solution Single Dose: One drop in the study administered one time
  One drop in the study administered one time in one day
Arm/Group | CBT-001 Ophthalmic Solution Single Dose
Number analyzed (Participants) | 24
participants
  Mild eye irritation | 3
  Mild foreign body sensation | 1

3. Secondary Outcome: Corneal Pterygium Lesion Length Change From Baseline
Description: The Corneal Pterygium Lesion Length is measured from digital images of the eye by an independent image reading center.
Time Frame: 4 weeks
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: mm
Groups:
- CBT-001 Ophthalmic Solution: One drop in the study administered three times daily (TID)
  CBT-001: One drop in the study administered three times daily (TID)
- Vehicle: One drop in the study administered three times daily (TID)
  Vehicle: One drop in the study administered three times daily (TID)
Arm/Group | CBT-001 Ophthalmic Solution | Vehicle
Number analyzed (Participants) | 25 | 23
mm | -0.11 (0.3) | 0.16 (0.36)
Statistical Analysis 1: Comparison: CBT-001 Ophthalmic Solution vs Vehicle; Test type: Superiority; p = 0.007, ANOVA; Mean Difference (Final Values) = 0.27

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CBT-001 Ophthalmic Solution Single Dose | Vehicle Multi-dose | CBT-001 Ophthalmic Solution Multi-dose
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/25 | 0/26
Other Adverse Events (participants affected / at risk) | 4/24 | 2/25 | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-001 Ophthalmic Solution Single Dose (N=24) | Vehicle Multi-dose (N=25) | CBT-001 Ophthalmic Solution Multi-dose (N=26)
Transient ischaemic attack (Blood and lymphatic system disorders) | NA | 1 (1) | 0 (0) — not treatment related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-001 Ophthalmic Solution Single Dose (N=24) | Vehicle Multi-dose (N=25) | CBT-001 Ophthalmic Solution Multi-dose (N=26)
Conjunctival Discoloration (Eye disorders) | 0 (0) | 0 (0) | 14
Foreign Body Sensation in Eyes (Eye disorders) | 1 (1) | 0 | 2
Lacrimation Increased (Eye disorders) | 0 (0) | 0 | 2
Dysgeusia (General disorders) | 0 (0) | 0 | 2
Influenza A infection (Infections and infestations) | 0 (0) | 2 | 0
Eye irritation (Eye disorders) | 3 (3) | 0 (0) | 0 (0) — Mild eye irritation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT03049852/Prot_SAP_000.pdf